CLINICAL TRIAL: NCT02684656
Title: Pilot Study of Lowering Plasma Oxalate With Hemodiafiltration to Reduce Systemic Inflammation in Patients With End-Stage Renal Disease (ESRD)
Brief Title: Reduction of Oxalate and Inflammation by Hemodiafiltration vs. Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: Renal Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: UErlangen-Nurnberg
Record Dates: First submitted 2016-02-09; First posted 2016-02-18 (Estimated); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Chronic Kidney Disease Requiring Chronic Dialysis
Keywords: Oxalate; Inflammation; Hemodiafiltration; Hemodialysis; Oxalate Blood Sample
MeSH Terms: conditions — Inflammation | interventions — Renal Dialysis; Hemodiafiltration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hemodialysis (Active Comparator): Intervention: Patients will be switch to hemodialysis and basal plasma oxalate levels as well as oxalate removal by hemodialysis will be determined after two weeks of treatment.
  Interventions: Procedure: Hemodialysis
- Hemodiafiltration (Active Comparator): Intervention: Patients will be switch back to hemodiafiltration and basal plasma oxalate levels as well as oxalate removal by hemodiafiltration will be determined after two weeks of treatment.
  Interventions: Procedure: Hemodiafiltration

INTERVENTIONS:
Procedure: Hemodialysis — Hemodialysis >/=4h
  Arms: Hemodialysis
Procedure: Hemodiafiltration — Hemodiafiltration >/=4h, > 20l convection
  Arms: Hemodiafiltration

SUMMARY:
The health care burden of CKD is substantial and growing with 10-15% of the population affected in both developed and developing countries. It is well established that CKD is associated with systemic inflammation, which promotes cardiovascular disease and body wasting. However, causal therapies to treat systemic inflammation, and treat its adverse consequences remain sparse. As kidney function declines in all forms of CKD, oxalate levels increase in the plasma, leading to increased systemic exposure to oxalate and consequent tissue injury. Work from the investigators has shown that elevated plasma oxalate levels activate the NLRP3 inflammasome which in turn leads to the processing and release of cytokines. The investigators seek to test the hypothesis that oxalate contributes to the systemic inflammation observed in patients with end-stage renal disease (ESRD). The investigators plan to define the association between plasma oxalate levels and signs of systemic inflammation in patients on hemodialysis. In a second step the investigators will examine whether hemodiafiltration lowers plasma oxalate more efficiently than hemodialysis and reduces signs of systemic inflammation. Confirmation of the hypothesis may lead to the identification of oxalate as a novel therapeutic target for interventional trials aimed at reducing plasma oxalate in patients with ESRD.

DETAILED DESCRIPTION:
The positive interaction between diffusive and convective flux has suggested that hemodiafiltration (HDF) has a higher oxalate extraction rate as compared with hemodialysis (HD). However, it has not been evaluated whether HDF can lower predialysis oxalate levels below the level of supersaturation. By using an intra-individual approach with the inclusion/exclusion criteria listed for the study, we plan to determine plasma oxalate and cytokine levels in 20 patients (10 on regular duration HD, 10 patients on extended duration HD) before dialysis. Subsequently, patients will be switched to HDF and plasma oxalate concentration and cytokines will be analyzed again two weeks following HDF treatment. Plasma oxalate (Pox) will be measured at beginning of treatment, mid, end and 2 hrs post treatment (to determine rebound) in order to provide oxalate kinetics on HD/HDF treatment. Cytokines will only be measured pre HD/HDF treatment to assess steady state inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Blood Flow ≥ 250 ml/min
* Dialysate Flow ≥ 500 ml/min
* Urinary Excretion < 400 ml/24h
* Duration of Dialysis ≥ 4h
* On HDF/HD treatment for ≥ 4 weeks
* Extended HDF/HD for ≥ 4 weeks

Exclusion Criteria:

* Recirculation (online measurement) > 15%
* Single needle dialysis or single lumen catheter
* Substitution volume of < 20l on HDF

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Plasma oxalate | 6 months

SECONDARY OUTCOMES:
Cytokines measured by multiplex analysis | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Felix Knauf, MD, Principal Investigator — University Erlangen-Nuremberg, Germany; Kai-Uwe Eckardt, MD, Principal Investigator — University Erlangen-Nuremberg, Germany; Fred Finkelstein, MD, Principal Investigator — Medical Director of New Haven Home Dialysis; Peter S Aronson, MD, Principal Investigator — Yale University New Haven, USA; Chirag Parikh, MD, Principal Investigator — Yale University New Haven; Mark A Perazella, MD, Principal Investigator — Yale University New Haven
Locations (1):
- Nephrology Department, University Hospital Erlangen, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoppe B, Kemper MJ, Bokenkamp A, Portale AA, Cohn RA, Langman CB. Plasma calcium oxalate supersaturation in children with primary hyperoxaluria and end-stage renal failure. Kidney Int. 1999 Jul;56(1):268-74. doi: 10.1046/j.1523-1755.1999.00546.x. PMID 10411702
- [Background] Knauf F, Asplin JR, Granja I, Schmidt IM, Moeckel GW, David RJ, Flavell RA, Aronson PS. NALP3-mediated inflammation is a principal cause of progressive renal failure in oxalate nephropathy. Kidney Int. 2013 Nov;84(5):895-901. doi: 10.1038/ki.2013.207. Epub 2013 Jun 5. PMID 23739234